CLINICAL TRIAL: NCT04763395
Title: Liver Function Test Abnormalities in COVID-19 Egyptian Patients
Brief Title: Liver Function Test Abnormalities in COVID-19
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mona Mohammed Abdelrhman, Principal investigator, Sohag University
Other Study IDs: Soh-Med-21-02-27
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Liver Function Tests Abnormalities
Keywords: Liver function tests; Covid19; Severity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-severe COVID19: * Patients with mild symptoms (i.e., fever, cough, expectoration, and other upper respiratory tract symptoms), and without abnormalities, or with mild changes on chest radiography, were classified as non-severe types.
  * A mild change in chest radiography is defined by multiple small patchy shadows and interstitial changes, mainly in the outer zone of the lung and under the pleura.
  Interventions: Other: No intervention
- Severe Covid19: Severe COVID19 was defined by the presence of any of the following conditions: i) significantly increased respiration rate (RR): RR >-30 times/minute; ii) hypoxia: oxygen saturation (resting state) <-93%; iii) blood gas analysis: partial pressure of oxygen/fraction of inspired oxygen (PaO2) /FiO2) <- 300 mmHg (millimeters of Mercury), or iv) the occurrence of respiratory or another organ failure that require Intensive care unit (ICU) monitoring and treatment, or shock
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
With the increasing number of COVID-19 infected patients, several studies reported that the liver is the most frequently affected organ after lung damage. The percentage of infected patients who had abnormal levels of transaminases (alanine aminotransferase (ALT) and aspartate aminotransferase (AST)) was about 14.8-53.1%. The elevation in serum bilirubin was mostly mild.

Aims of work:

* To study liver function tests abnormalities in Egyptian patients who infected with COVID19
* To evaluate if liver function test abnormalities are related to the severity of the Covid19.

DETAILED DESCRIPTION:
This retrospective study will be conducted on 100 patients who were diagnosed as SARS COVID19 positive. The data will be collected from patient records in COVID19 isolation hospitals in Sohag governorate and isolation department in Sohag university hospitals during the period from the start of June 2020 to the end of July 2020.

The study protocol will be approved by the Scientific Research Ethical Committee, Faculty of Medicine, Sohag University.

Inclusion criteria:

Patients with Covid19 positive PCR.

Exclusion Criteria:

Patients with chronic liver diseases as liver cirrhosis, Hbs Ag positive, or patients having anti-HCV antibodies positive and HCV RNA positive.

The Data will be collected according to the rules of the Sohag university ethical committee. The following will be collected

1. Data about clinical manifestations including fever, cough, dyspnea, fatigue, and diarrhea.
2. Laboratory investigation:

   * CBC -Total bilirubin and direct
   * AST - ALT
   * Albumin - Prothrombin time and concentration
   * CRP -D-dimer
   * Serum ferritin
3. Assessment of the severity of the disease:

Patients were classified into severe or mild cases based on results from chest radiography, clinical examination, and symptoms.

* Patients with mild symptoms (i.e., fever, cough, expectoration, and other upper respiratory tract symptoms), and without abnormalities, or with mild changes on chest radiography, were classified as non-severe types.
* A mild change in chest radiography is defined by multiple small patchy shadows and interstitial changes, mainly in the outer zone of the lung and under the pleura.
* Severe pneumonia was defined by the presence of any of the following conditions: i) significantly increased respiration rate (RR): RR >-30 times/minute; ii) hypoxia: oxygen saturation (resting state) <-93%; iii) blood gas analysis: partial pressure of oxygen/fraction of inspired oxygen (PaO2) /FiO2) <- 300 mmHg (millimeters of Mercury), or iv) the occurrence of respiratory or another organ failure that require Intensive care unit (ICU) monitoring and treatment, or shock

  4. Statistical analysis: Data will be analyzed using STATA version 14.2 (Statistical Software: Release 14.2 College Station, TX: Stata Corp LP). Quantitative data will be represented as mean, standard deviation, median and range. normally distributed. Qualitative data will be presented as numbers and percentages. Chi square test will be used for comparison of percentages in different groups. P value will be considered significant if it was less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

Patients with Covid19 positive PCR.

Exclusion Criteria:

Patients with chronic liver diseases as liver cirrhosis, Hbs Ag positive, or patients having anti-HCV antibodies positive and HCV RNA positive

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients who were diagnosed as SARS COVID19 positive. The data will be collected from patient records in COVID19 isolation hospitals in Sohag governorate and isolation department in Sohag university hospitals during the period from the start of June 2020 to the end of July 2020
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Percentage of liver function tests abnormalities in Egyptian patients who infected with COVID19 -To evaluate if liver function test abnormalities are related to the severity of the Covid19. | during the period from the start of June 2020 to the end of July 2020
Risk factors of Liver function test abnormalities | during the period from the start of June 2020 to the end of July 2020
Liver function test abnormalities among patients with severe and non-severe disease | during the period from the start of June 2020 to the end of July 2020

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Mahmoud, lecturer, Study Chair — Sohag University; Mustafa Younis, lecturer, Study Chair — Sohag University; Mahmoud Mahmoud, lecturer, Study Chair — Sohag University
Locations (1):
- Mona Mohammed Abdelrhman, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lai CC, Shih TP, Ko WC, Tang HJ, Hsueh PR. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and coronavirus disease-2019 (COVID-19): The epidemic and the challenges. Int J Antimicrob Agents. 2020 Mar;55(3):105924. doi: 10.1016/j.ijantimicag.2020.105924. Epub 2020 Feb 17. PMID 32081636
- [Background] Mao R, Liang J, Shen J, Ghosh S, Zhu LR, Yang H, Wu KC, Chen MH; Chinese Society of IBD, Chinese Elite IBD Union; Chinese IBD Quality Care Evaluation Center Committee. Implications of COVID-19 for patients with pre-existing digestive diseases. Lancet Gastroenterol Hepatol. 2020 May;5(5):425-427. doi: 10.1016/S2468-1253(20)30076-5. Epub 2020 Mar 11. No abstract available. PMID 32171057
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Zhang C, Shi L, Wang FS. Liver injury in COVID-19: management and challenges. Lancet Gastroenterol Hepatol. 2020 May;5(5):428-430. doi: 10.1016/S2468-1253(20)30057-1. Epub 2020 Mar 4. No abstract available. PMID 32145190